CLINICAL TRIAL: NCT06291298
Title: COGMUSE-AUT: Novel Adaptive Cognitive Training in Autistic Adults with Co-occurring Insomnia
Brief Title: Novel Adaptive Cognitive Training in Autistic Adults with Co-occurring Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Ashley Curtis, Assistant Professor, University of South Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY006542
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder; Insomnia
MeSH Terms: conditions — Autism Spectrum Disorder; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Pilot test COGMUSE-AUT in a small sample of autistic adults with co-occurring insomnia on primary and secondary outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- COGMUSE-AUT (Experimental): Participants will complete the computerized cognitive training intervention for 60 minutes per day, 3 times per week for 6 weeks at home totaling to 18 hours.
  Interventions: Behavioral: COGMUSE-AUT

INTERVENTIONS:
Behavioral: COGMUSE-AUT — The computerized training exercises and brain games help stimulate cognitive functions while providing real-time monitoring on the evolution of participants' skills.

SUMMARY:
The proposed study will test the usability and feasibility of a novel cognitive training (COGMUSE) for autistic adults with co-occurring insomnia (COGMUSE- AUT). Participants (n=15) will complete the cognitive training intervention for 60 minutes per day, 3 times per week for 6 weeks at home totaling to 18 hours. Weekly check-ins will be conducted by study staff over Teams to ensure adherence to the treatment and provide an opportunity for qualitative feedback on the game sessions played. During these 6 weeks, participants will fill out daily (2x/day) electronic sleep diaries and wear an actigraph device (GENEActiv). GENEActiv is a watch-like device that monitors light and movement activity.

ELIGIBILITY:
Inclusion Criteria:

1. 18+ years of age
2. Diagnosed with ASD (see 2a).
3. Verbal IQ >= 70 (Measured via the Weschler Abbreviated Scale of Intelligence 2nd Edition28); to ensure verbal skills sufficient to participate in treatment
4. Able to undergo actigraphy assessment
5. Can read and understand English
6. Diagnosed with insomnia (See 3a).
7. No prescribed or OTC sleep medications for 1+ month, or stabilized on medications for 6+ weeks.

2a) ASDb: a) previous DSM diagnosis of ASD (self-reported by ASD adult and guardian; confirmed by clinical documentation provided to project coordinator), 2) evaluation using gold-standard diagnostic tools (i.e., Autism Diagnostic Observation Schedule (ADOS) and/or Autism Diagnostic Interview -Revised [ADI-R]).

3a) Insomnia: a) insomnia complaints for 6+ months that b) occur despite adequate opportunity and circumstances for sleep, c) consist of 1 or more of the following: difficulty falling asleep, staying asleep, or waking up too early, d) daytime dysfunction (mood, cognitive, social, occupational) due to insomnia, f) baseline diaries and actigraphy indicate >30 minutes of sleep onset latency or wake after sleep onset on 6 or more nights.

Exclusion Criteria:

1. unable to provide informed consent
2. diagnosis of sleep disorder other than insomnia [i.e., sleep apnea (apnea/hypopnea index, AHI >15), Periodic Limb Movement Disorder (myoclonus arousals per hour >15)],
3. comorbid bipolar or seizure disorder (due to risk of sleep restriction treatment)
4. other major psychopathology except depression or anxiety (e.g., suicidal ideation/intent, psychotic disorders)
5. severe untreated psychiatric comorbidity
6. psychotropic or other medications (e.g., beta-blockers) that alter sleep
7. participation in non-pharmacological treatment (including CBT) for pain, sleep or mood outside current trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Objective Cognition-National Institute of Health Toolbox | Up to 10 weeks
  A computerized cognitive test battery measuring performance across several domains:
  executive function (Flanker inhibitory control task), Dimensional Card Sort Test (measures cognitive flexibility, accuracy score), working memory (List Sorting Task), verbal (episodic) memory (Auditory Verbal Learning Task) will be administered.

SECONDARY OUTCOMES:
Objective Slee-Daily Actigraphy | Up to 10 weeks
  GENEActiv (Activiinsights), a watch-like device that monitors light and gross motor activity, will be worn 24 hours/7 days for 2 weeks at each assessment point.
Subjective Sleep- Electronic Daily Sleep Diaries | Up to 10 weeks
  Online diaries completed each morning (~5 mins) during 2-week assessment periods and 6 weeks training. Variables: sleep onset latency (time from lights-out until sleep onset), wake time after sleep onset, sleep efficiency (% time spent sleeping while in bed).
Insomnia Severity Index | Up to 10 weeks
  5-item survey completed by adult with autism and parent/guardian if needed. Brief measure of current perception of insomnia symptom severity, distress and daytime impairment. Commonly used in insomnia treatment outcome research.
Sleep Habits Questionnaire | Up to 10 weeks
  Modified Sleep Habits Questionnaire, based on child version and modified for adults. This questionnaire gauges sleep habits and possible difficulties with sleep.
Pre-Sleep Arousal | Up to 10 weeks
  -Pre-sleep Arousal Scale is a 16-item self-report questionnaire comprising both cognitive and somatic manifestations of arousal. This questionnaire will be completed by autistic adult with assistance from parent/guardian as needed.
WHO Quality of Life-BREF | Up to 10 weeks
  This measure assesses quality of life (QOL) within the context of an individual's culture, value systems, personal goals, standards and concerns.
Mood | Up to 10 weeks
  State-Trait Anxiety Inventory: Inventory that asks respondents to rate how true 20 self-descriptive statements (e.g., I feel calm) are on a 4-point scale (1 = not at all, 4 = very much so). Typically, respondents are asked to rate statements according to how they generally feel (trait-anxiety scale) and how they feel in the current moment (state-anxiety scale). Total scores range from 20 to 80, with higher scores indicating greater maladjustment.
Depression | Up to 10 weeks
  - Beck Depression Inventory (II): 21-item inventory that asks respondents to rate on a scale of 0 (no depressive feelings) to 3 (most depressive feelings) their feelings towards various aspects of daily living/situations. Higher total scores indicate worse depressive symptoms.
Adaptive Behavior Assessment System (ABAS-III) | Up to 10 weeks
  Adaptive functioning --This assessment measures behaviors suitable for adults displayed in several domains such as communication, community use, functional academics, home living, health and safety, leisure, self-care, self-direction, social, and work. The assessment will be filled by the adult with autism with the help of the caregiver if necessary. Answers are provided in a likert scale with 0=is not able to do this behavior to 3= always (or almost always).
Game-related experience (completed during intervention) | Up to 10 weeks
  Sessions played -- The graduate research assistant will check adherence through an online portal storing COGMUSESM data during weekly Teams check-ins with participant. Participants will also provide qualitative feedback on the game sessions played.
  Weekly game -- Maximum test scores recorded.
  Game Engagement Questionnaire - Completed at the end of intervention; Participants rate from 0 (none) to 4 (extremely) the degree to which they agree with 33 aspects of game experiences. Total score measures game engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley F Curtis, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No